CLINICAL TRIAL: NCT02891551
Title: A Non-interventional Observational Post Authorization Study to Evaluate Safety and Efficacy in Patients Receiving Azacitidine in Daily Clinical Practice in the Netherlands (OCEAN)
Brief Title: An Observational Post Authorisation Study to Evaluate Safety and Efficacy in Patients Receiving Azacitidine in Daily Clinical Practice in the Netherlands
Acronym: OCEAN
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-VZ-NL-001
Record Dates: First submitted 2015-10-20; First posted 2016-09-07 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute
Keywords: Leukemia; Chronic; Acute; Observational; Non-interventional; OCEAN; Netherlands; azacitidine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Leukemia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving Azacitidine per daily clinical practice

SUMMARY:
The study design is a prospective, non-interventional, observational single arm study.

A minimum of 150 patients will be recruited from approximately 30 haematology/oncology sites in the Netherlands. In all cases, the decision to treat the patient with azacitidine was already made prior to the decision to enter the subject into the study.

Recruitment will continue until end of June 2015, provided a minimum of 150 patients have been included in the study. When this date is reached, all patients on azacitidine will continue to be followed until the last patient enrolled has been followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who understand and voluntarily sign an informed consent form.
* Patients who are treated with azacitidine in accordance with registered indication and clinical practice.

Exclusion Criteria:

* Refusal to participate in the study.
* Participation in an interventional clinical study.
* Patients previously treated with azacitidine except when given as induction therapy for a maximum of three courses.
* Women who are pregnant or breast-feeding.
* Hypersensitivity to the active substance or to any of the excipients.
* Advanced malignant hepatic tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who are treated with azacitidine in accordance with registered indication and clinical practice. In all cases, the decision to treat the patient with azacitidine was already made prior to the decision to enter the subject into the study
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 4 years
  Adverse events will be classified using the Medical Drug Regulatory Activities (MedDRA) classification system. The severity of the toxicities will be graded according to the NCI CTCAE VERSION 4.03 whenever possible

SECONDARY OUTCOMES:
Fact-Anemia Quality of life questionnaire | Up to approximately 4 years
  The Functional Assessment of Cancer Therapy-Anemia (FACT-An) questionnaire was used to assess health-related quality of life (HRQoL). In addition to general HRQoL, the FACT-An measures the impact of fatigue and other anemia-related symptoms on patient functioning.
Percentage of patients with a Haematological Response in daily clinical practice using the International Work Group Criteria in Myelodysplastic Syndrome Assessed by the Investigator | Up to approximately 4 years
  Hematologic Response according to the 2000 International Working Group (IWG) response criteria for Myelodysplastic Syndrome (MDS)
Percentage of patients with a Hematologic Improvement Using International Working Group (IWG Criteria for Hematologic Improvement Cheson 2000) Criteria for Myelodysplastic Syndrome (MDS) and Assessed by the investigator in daily clinical practice | Up to approximately 4 years
  Overall hematological improvement (HI) was defined as any type (major or minor) of improvement of HI-E, HI-P, or HI-N. Criteria: Pretreatment=hemoglobin <100g/L or RBC transfusion-dependent, platelet count <100x10^9/L or platelet transfusion dependent, absolute neutrophil count <1.5x10^9/L. Sponsor's determination was derived using clinically relevant data.
  Denominator for progression/relapse after HI included participants who had achieved HI.
Time to treatment Failure daily clinical practice | Up to approximately 4 years
  Time to Treatment Failure is defined as the time from randomization to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death.
Overall Survival in daily clinical practice | Up to approximately 4 years
  Overall survival (OS) was assessed using the time between randomization and the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Jan Koedam, MSc, Study Director — Celgene